CLINICAL TRIAL: NCT02048189
Title: Treatment With Continuous Sub-cutaneous Insulin Infusion Via a Portable Pump Versus Discontinuous Insulin Infusion Via Multiple-injections in Type 2 Diabetes: Study of Insulin Sensitivity in the 2 Types of Treatment
Brief Title: Treatment With Continuous Sub-cutaneous Insulin Infusion Via a Portable Pump Versus Discontinuous Insulin Infusion Via Multiple-injections in Type 2 Diabetes
Acronym: TRICIDIA
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: recruitment difficulties
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RUDONI PARI 2011
Record Dates: First submitted 2014-01-23; First posted 2014-01-29 (Estimated); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Patient With Type 2 Diabetes Treated With Insulin Using a Baseline/Bolus Strategy
MeSH Terms: interventions — Insulin Detemir; insulin glulisine

ARMS (2):
- Intensified multiple injections (Other)
  Interventions: Drug: LEVEMIR
- Pumps (Other)
  Interventions: Drug: APIDRA

INTERVENTIONS:
Drug: LEVEMIR
  Arms: Intensified multiple injections
Drug: APIDRA
  Arms: Pumps

SUMMARY:
This is an open multicentre, randomized study to compare two treatment arms. One arm called "intensification of multiple injections" in which the patient will receive one supplementary injection of LEVEMIR®: that is to say 5 injections per day, and an arm called "continuous insulin infusion" via an external pump with APIDRA®.

In the pump arm: a favorable effect in terms of improved insulin sensitivity, improved metabolic equilibrium, a decrease in the area under the baseline and prandial hyperglycemia curve noted during the continuous glycemia recording; an improvement in quality of life compared with treatment using multiple injections.

ELIGIBILITY:
Inclusion Criteria:

* Persons who have provided written informed consent
* Age > 18 years
* Patients with type 2 diabetes treated with insulin using a basal / bolus strategy for at least 6 months
* Doses of insulin > 0.7 U / Kg / d
* HbA1c ≥ 7.5 %
* Without OAD for at least 4 weeks (sulfamides, Incretines, glinides, acarbose) except Metformin
* BMI ≥ 28.5 kg / m2
* Diabetes diagnosed for at least 10 years
* Patients able to monitor themselves and manage an insulin pump.

Exclusion Criteria:

* Patients treated with glitazones during the 3 months preceding inclusion
* Patients with proliferative ischemic retinopathy not treated by laser
* BMI < 28.5 kg / m2
* Presence of implantable material ( CI MRI )
* Pacemaker ( CI MRI )
* Pregnancy, breast feeding
* Medically significant physical or psychiatric inability, patients under guardianship or wards of court
* The practice of violent sports
* Poor conditions of hygiene
* Professional environment of extreme cold or heat.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-03-08 (Actual); Primary Completion 2015-02-26 (Actual)

PRIMARY OUTCOMES:
Mixed measurement of insulin secretion and insulin resistance | Change from baseline insulin secretion and insuline resistance at 6 month after starting the treatment

SECONDARY OUTCOMES:
Decrease in the time spent in baseline and prandial hyperglycemia | During the 6 months following initiation of the treatment

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU de Besancon, Besançon
  - CHU de Dijon, Dijon